CLINICAL TRIAL: NCT03959709
Title: A Randomized Controlled Trial Comparing the Pre-pectoral Versus Sub-pectoral Implant Placement in Immediate Breast Reconstruction
Brief Title: Pre-pectoral Versus Sub-pectoral Implant Placement in Immediate Breast Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1449
Record Dates: First submitted 2019-05-10; First posted 2019-05-22 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Mastectomy; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prepectoral implant placement (Experimental): Immediate acellular dermal matrix-assisted implant-based breast reconstruction with prepectoral implant placement.
  Interventions: Procedure: immediate acellular dermal matrix-assisted implant-based breast reconstruction with prepectoral implant placement.
- Subpectoral implant placement (Active Comparator): Immediate acellular dermal matrix-assisted implant-based breast reconstruction with subpectoral implant placement.
  Interventions: Procedure: Immediate acellular dermal matrix-assisted implant-based breast reconstruction with subpectoral implant placement

INTERVENTIONS:
Procedure: immediate acellular dermal matrix-assisted implant-based breast reconstruction with prepectoral implant placement. — On the day of surgery, after the completion of the mastectomy, the vascularity of the mastectomy flaps will be evaluated, and debridement is performed where necessary. A temporary implant sizer is placed in the pocket to assess the position and shape of the prepectoral pocket. The pocket is adjusted where necessary. A sheet of ADM (DermAcell) is then selected. The DermAcell will be prepared as per the manufacture's instructions and fenestrated using size 11 blade. The DermACELL piece will be trimmed to the appropriate shape and sutured to the superior medial and lateral edges of the pectoralis major muscle. The inferior edge will be sutured to the fascia at the level of the inframammary fold. Two closed suction drains will be placed (one below the mastectomy skin flap, and one below DermACELL). The implant will be inserted to the pre-pectoral pocket and several anchor sutures will be used to secure the superior-medial edge of DermACELL to mastectomy flap.
  Arms: Prepectoral implant placement
Procedure: Immediate acellular dermal matrix-assisted implant-based breast reconstruction with subpectoral implant placement — On the day of surgery, after the completion of the mastectomy, the vascularity of the mastectomy flaps will be evaluated, and debridement is performed where necessary. The reconstructive operative procedure will then proceeded with (1) elevation of the pectoralis major muscle with release of inferior attachments; (2) placement of implant subpectorally; (3) placement and suturing of DermACELL to constitute the inferolateral breast pocket; (4) placement of two closed suction drains (one superiorly between the pectoralis major and skin, and one inferiorly between the DermACELL and skin); (5) removal of sizer and placement of permanent to the pocket and (6) suture the inferior edge of DermACELL to the inferior edge of the pectoral major muscle. The skin will be closed and the dressing will be applied as standard protocol.
  Arms: Subpectoral implant placement

SUMMARY:
Despite the popularity and proved safety of prepectoral implant-based reconstruction, there is little evidence on long-term results and variables which could influence surgical outcome. So far, no specific guidelines or indications have been developed for prepectoral technique and heterogeneous inclusion criteria had been used in previous reports. There is a lack of studies documenting outcomes following ADM-assisted prepectoral breast reconstruction, and there are no randomised controlled trial studies that drawing a direct comparison of clinical or patient-reported outcomes between subpectoral and prepectoral groups.

The investigators hypothesized that immediate acellular dermal matrix-assisted implant-based breast reconstruction with prepectoral implant placement would result in less early postoperative pain but more reported implant rippling, requirement of more fat grafting and an equitable safety profile compared with ADM-assisted implant-based breast reconstruction with subpectoral implant placement.

The aim of this study is to evaluate the postsurgical pain, complications and patient-reported outcomes of prepectoral breast reconstruction versus subpectoral implant placement in immediate breast reconstruction.

DETAILED DESCRIPTION:
The investigators will employ a single centre RCT with duration of two years (July 1, 2019 - June 30, 2021). Participant recruitment and enrolment will occur at the Women's Health Center for 1 year (July 1, 2019 to June 30, 2020), followed by one year (June 30, 2021) of follow-up data collection, data analyses and dissemination.

At the preoperative consultation, the surgeon will determine if the patient is eligible for implant-based immediate reconstruction, using the inclusion and exclusion criteria.

A total of 56 patients or 23 patients per arm will be recruited. Randomization will be accomplished using randomly permuted blocks, and the randomization list will be prepared by a biostatistician with no clinical involvement in this trial. Randomization will be stratified on the basis of center and laterality of reconstruction (i.e., unilateral versus bilateral reconstruction).

The allocation sequence will be concealed by placing each randomization assignment in a sequentially numbered, opaque, sealed envelope. Consecutive envelopes will be delivered to the operating room by the on-site research study assistant once the mastectomy is complete. To prevent subversion of the allocation sequence, envelopes will not be opened until the attending surgeon confirms the absence of significant mastectomy flap necrosis and the fact that the patient does not undergo a concurrent axillary lymph node dissection.

All patients will be blinded to their treatment arm. Once the treatment arm is revealed, the attending surgeon will advise the surgical team (surgical assistants and operating room nurses) the surgical plan. While the surgical team will be aware of the randomization code, the rest of the postoperative care team (including recovery room staff, day surgery nursing staff, and clinic staff during follow-up visit), outcome assessors, and data analysts will be kept blinded to the intervention performed.

Outcome measures:

At the baseline visit, following informed consent, demographic data (age, BMI, laterality and comorbidities) will be collected. The participant will then complete the following questionnaires: Pre-operative Breast-Q™: The Breast-Q™ Reconstruction Module is a validated PRO developed specifically for patients undergoing breast reconstruction. The questionnaire evaluates patient-reported satisfaction, psychosocial, physical and sexual quality of life [1] Primary outcome: Postoperative Pain scores and 24-hour narcotic consumption Secondary outcomes: All outcomes are measured within or at 12 months of the initial surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female patient
* Ages 20-80
* All patients undergoing mastectomy for breast cancer or prophylaxis for breast cancer with immediate implant-based reconstruction
* Able to provide informed consent

Exclusion Criteria:

* Patients who have had prior chest wall or irradiation on the reconstructed side
* Patients not undergoing immediate breast reconstruction at the time of mastectomy
* Any patient with a contraindication to immediate breast reconstruction.
* Patients with history of smoking, BMI> 40, and D cup breast size or grade III ptosis are all contraindications to immediate breast reconstruction as the risk of postoperative complications are significantly higher (wound infection, dehiscence, implant loss, seroma) than the average patient and thus these patients would be excluded from the study.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 56 (Estimated)
Dates: Start 2019-08-22 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain and 24-hour narcotic consumption | 24 hours
  Postoperative Pain will be scored using Numerical rating scale. The scale ranges from 0 to 10 indicating the level of pain. Zero indicates the absence of pain, while 10 represents the most intense pain (no pain = 0, mild = 1-3, moderate = 4-6, severe = 7-10).

SECONDARY OUTCOMES:
Mastectomy flap necrosis | 4 weeks
  Skin loss of mastectomy flap
Rate of seroma | 4 weeks
  Episodes of seroma formation requiring aspiration
Rate of infection | 3 months
  Cellulitis and abscess
Rate of Explantation | 1 year
  Loss of implant
Number of Revisional surgeries | 1 year
  return to operating room for more surgeries
Rate of Wound | 3 months
  incision dehiscence or debridement
Rate of Capsular contracture | 1 year
  Tightening, firmness and pain of reconstructive breast
BREAST-Q© Pre-operative scale | Before Surgery
  The BREAST-Q© modules is comprised of the following two overarching themes (or domains): 1) Health-Related Quality of Life (QOL) and 2) Patient Satisfaction. Under each of these domains, there are six subthemes; QOL: 1) Psychosocial, 2) Physical and 3) Sexual well-being; and Patient Satisfaction: 4) Satisfaction with Breasts, 5) Satisfaction with Outcome and 6) Satisfaction with Care. Body image is an important concept for breast surgery patients. Preoperative scales: Satisfaction with Breasts, Psychosocial, Sexual and Physical Well-being Chest
  There is no overall or total BREAST-Q© score, only scores for each independent scale. All BREAST-Q© scales are transformed into scores that range from 0-100. The scores are computed by adding the response items together and then converting the raw sum scale score to a score from 0-100. For all BREAST-Q© scales, a higher score means greater satisfaction or better QOL (depending on the scale). The score is from 0 (worst) to 100 (best).
BREAST-Q© Post-operative | 3 months and 12 months
  The BREAST-Q© modules is comprised of the following two overarching themes (or domains): 1) Health-Related Quality of Life (QOL) and 2) Patient Satisfaction. Under each of these domains, there are six subthemes; QOL: 1) Psychosocial, 2) Physical and 3) Sexual well-being; and Patient Satisfaction: 4) Satisfaction with Breasts, 5) Satisfaction with Outcome and 6) Satisfaction with Care. Body image is an important concept for breast surgery patients.
  Postoperative scales: Satisfaction with Doctor, Medical Team and Office Staff
  There is no overall or total BREAST-Q© score, only scores for each independent scale. All BREAST-Q© scales are transformed into scores that range from 0-100. The scores are computed by adding the response items together and then converting the raw sum scale score to a score from 0-100. For all BREAST-Q© scales, a higher score means greater satisfaction or better QOL (depending on the scale).
  The score is from 0 (worst) to 100 (best).

CONTACTS AND LOCATIONS:
Overall Officials: Jing Zhang, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No